CLINICAL TRIAL: NCT06533735
Title: Parent Web - Support for Families With Young People
Acronym: PWS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Laura Ferrer Wreder, Associate Professor of Psychology, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FoUI-993293
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Family Conflict; Family Relations; Family Dysfunction
Keywords: parent training; universal; youth externalizing problems; family conflict; warmth in families

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled experiment (RCT) with a wait-list control group
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Immediate Intervention Group (Experimental): The immediate intervention group will take part in the online parent training program called the Parent Web (PW), with pre and post testing (before and after intervention).
  Interventions: Behavioral: Parent Web
- Wait-List Control Group (Other): This is a group of parents who are in a wait-list control group and will receive the Parent Web, after pre and post testing.
  Interventions: Behavioral: Parent Web

INTERVENTIONS:
Behavioral: Parent Web — Parent-Web (PW) is internet delivered and rooted in social learning and coercion theory, PW supports parenting practices and parent-child interactions encouraging prosocial behavior and emotion regulation, reduce coercive parenting, improve communication, problem solving, and warmth. PW has a universal and selective edition. Universal PW has 5 basic modules (1 module per week, 6-8 weeks) and bonus modules. Basic modules contain information, exercises, and videos of actors showing parenting practices. A family guide supports parents through modules.

SUMMARY:
To test an online parent training program. Relative to a randomized wait-list control group, those in the Parent Web (PW) will show benefits on well-being, parenting, stress, youth mental health.

DETAILED DESCRIPTION:
Parent-Web (PW) is internet delivered parent education that is created and developed by researchers at Karolinska Institute's Department of Clinical Neuroscience, namely Kajsa Lönn-Rhodin, Martin Forster, and Pia Enebrink. An effectiveness trial of the universal edition of the Parent Web is made possible through a research collaboration with Pia Enebrink. PW is derived from social learning and coercion theory. PW aims to support parenting practices and parent-child interactions encourage prosocial behaviour and emotion regulation, reduce coercive parenting, improve communication, problem solving, and warmth within families. PW has a universal and selective edition. Universal PW has 5 basic modules (1 module per week, 6-8 weeks) and bonus modules. Basic modules contain information, exercises, and videos of actors showing parenting practices. A family guide supports PW participants through PW modules. This study will test the effects of universal PW with a general population derived sample of parents living in Region Stockholm. All PW trial participants are parents to at least one adolescent child who is aged 11-13 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have to be parents and/or legal guardians of at least one 11 to 13 year old child.
2. Participants must live in Region Stockholm.

Exclusion Criterion:

1. The target child (the 11 to 13-year-old) is presently receiving mental health treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in parent rating of child's emotional problems, conduct problems, hyperactivity, peer problems and prosocial behavior | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rating of their child's emotional problems, conduct problems, hyperactivity, peer problems and prosocial behavior as indexed by the Strengths and Difficulties Questionnaire (SDQ).
  The SDQ consists of 25 items rated on a 3-point Likert scale with response options that range from 0 = not true, 1 = somewhat true, 2 = certainly true. Higher scores indicate a worse outcome on the emotional problems, conduct problems, hyperactivity, peer problems scale scores. Higher scores on the prosocial behavior scale indicate a better outcome.
Change from baseline in parent rated view of their child's behavioral problems/defiant behavior | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent view of their child's behavioral problems/defiant behavior as measured by the Oppositional Defiant Scale of the Disruptive Disorder Rating Scale (DBD) which consists of 7 items rated on a 4-point scale ranging from 1 (not at all) to 4 (very much). Higher scores indicate a worse outcome.
Change from baseline in parent rated family warmth and conflict | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated warmth and conflict. Warmth and conflict are indexed by eight items rated on a five-point scale from 1 (never) to 5 (more than 7 times). Five items measure parent-child warmth and three items measure parent-child conflicts. Higher scores on parental warmth scale indicate a better outcome. Higher scores on the parent-child conflicts scale score indicate a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in parent rated encouragement of positive behaviors, setting limits, and proactive parenting behaviors | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated encouragement of positive behaviors, setting limits, and proactive parenting behaviors as indexed by the Parenting Children and Adolescents Scale (PARCA). The PARCA has 19 items rated on a five-point scale 1 = never to 5 = Very Often. The scale has three subscales on encouragement of positive behaviors, setting limits, and proactive parenting behaviors. Higher scores indicate a better outcome.
Change from baseline in parent rated stress | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated stress as measured by the Perceived Stress Scale (PSS). PSS consists of 10 questions about perceived stress during the last month rated on a 5-point Likert scale (0 = Never to 4 = Very Often). The scale measures the extent to which situations in one's life are assessed and perceived as stressful and current stress levels. Higher scores indicate a worse outcome.
Change from baseline in parent rated health | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated health as measured by the Hospital Anxiety and Depression Scale (HAD). HAD consists of two scales (a total of 14 items), one for anxiety and one for depression with seven questions each. Items are rated on a 4-point Likert scale. Higher scores indicate a worse outcome.
Change from baseline in parent rated parents validation of their child's emotions when expressed | [Time Frame: Immediate PW group pretest in Fall/Winter 2024. Post test up to 10 months after pretest. Wait-list group pretest in Fall/Winter 2024. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1]
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated affective style as measured by the tolerating subscale of the Affective Style Questionnaire (ASQ). The ASQ consists of five items (rated on a 3 point Likert scale,
  1 = Completely Agree to 3 = Completely Disagree) that examine how parents view their own validation of their child's emotions when expressed. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The datasets to be collected in this trial are not readily available because this study's ethical review does not allow for study data to be in a public repository. For meta-analysis or confirmation of published study results, individual level, de-identified data requests will be reviewed when made by qualified researchers (e.g., Ph.D.) along with ethical permission under Swedish law regarding secondary data analysis. Requests to access the datasets should be directed to Laura Ferrer-Wreder (laura.ferrer-wreder@psychology.su.se)

REFERENCES:
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Malmberg M, Rydell AM, Smedje H. Validity of the Swedish version of the Strengths and Difficulties Questionnaire (SDQ-Swe). Nord J Psychiatry. 2003;57(5):357-63. doi: 10.1080/08039480310002697. PMID 14522609
- [Background] Pelham WE Jr, Gnagy EM, Greenslade KE, Milich R. Teacher ratings of DSM-III-R symptoms for the disruptive behavior disorders. J Am Acad Child Adolesc Psychiatry. 1992 Mar;31(2):210-8. doi: 10.1097/00004583-199203000-00006. PMID 1564021
- [Background] Criss MM, Shaw DS. Sibling relationships as contexts for delinquency training in low-income families. J Fam Psychol. 2005 Dec;19(4):592-600. doi: 10.1037/0893-3200.19.4.592. PMID 16402874
- [Background] Wetterborg D, Enebrink P, Lonn Rhodin K, Forster M, Risto E, Dahlstrom J, Forsberg K, Ghaderi A. A pilot randomized controlled trial of Internet-delivered parent training for parents of teenagers. J Fam Psychol. 2019 Oct;33(7):764-774. doi: 10.1037/fam0000541. Epub 2019 Jun 17. PMID 31204818
- [Background] Ringle JL, Mason WA, Oats RG, Cogua J. Parenting Children and Adolescents (PARCA) scale English to Spanish translation: An investigation of measurement invariance. J Fam Psychol. 2019 Dec;33(8):938-944. doi: 10.1037/fam0000559. Epub 2019 Jul 18. PMID 31318263
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Hofmann SG, Kashdan TB. The Affective Style Questionnaire: Development and Psychometric Properties. J Psychopathol Behav Assess. 2010 Jun 1;32(2):255-263. doi: 10.1007/s10862-009-9142-4. PMID 20495674